CLINICAL TRIAL: NCT01840670
Title: Influence of Central Venous and Abdominal Pressures on the Inferior Vena Cava Shape and Size
Brief Title: Central Venous and Abdominal Pressures and the Inferior Vena Cava
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Franco Cavaliere, Professor, Catholic University of the Sacred Heart
Other Study IDs: UCSC-123-FC
Record Dates: First submitted 2013-04-17; First posted 2013-04-26 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Hypovolemia
Keywords: Inferior Vena Cava; Central Venous Pressure; Abdominal Pressure
MeSH Terms: conditions — Hypovolemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Rapid fluid load test — The test will be performed by infusing 250-300 mL/m2 Body Surface Area of 6% hydroxyethyl starch 6% 130/0.4 (VoluvenR) in 30 minutes
  Other Names: VoluvenR

SUMMARY:
The elliptic shape of inferior vena cava (IVC) sections, while hindering the ultrasound measurement of IVC diameter, may provide a useful tool to estimate central venous pressure (CVP). Hypothetically, the higher is CVP and more the ratio R between minimum and maximum diameters approximates 1. The purpose of this study is to determine R values in four different sections before and after a fluid load test, in order to evaluate if R is affected by the test and at which level the variation is larger.

The secondary endpoint is to search for the parameter best predictive of the positivity of the fluid load test among IVC minimum and maximum diameters, eccentricity, section area, and blood velocity at the level that presented the largest variations after the fluid load.

DETAILED DESCRIPTION:
The study will be carried out during the first 6 hours after the end of cardiac surgery when patients are mechanically ventilated and sedated with propofol and remifentanil to achieve a Ramsey sedation score of 3-4. The following four steps will be carried out:

A) A baseline hemodynamic and ultrasound assessment with the head of the bed positioned at 30 °.

B) The measurement of abdominal pressure with the head of the bed placed in a horizontal position for 3 minutes.

C) A rapid fluid load test with the head of the bed raised again to be 30°. The test will be performed by infusing 250-300 mL/m2 Body Surface Area of 6% hydroxyethyl starch 6% 130/0.4 (VoluvenR) in 30 minutes and will be considered positive if the cardiac index increases by at least 15% above the baseline value.

D) A second hemodynamic and ultrasound assessment with the head of the bed positioned at 30 °.

Hemodynamic evaluation The hemodynamic assessment will be run out by evaluating heart rate, systemic arterial and pulmonary pressures, central venous pressure, and pulmonary wedge pressure. Cardiac output will be measured by the thermodilution technique; the mean of three measures will be taken; then cardiac index will be calculated by dividing the cardiac output by the body surface area.

Ultrasound measurements

IVC maximum and minimum diameters (which will be defined as anteroposterior and lateral) will be measured at the end of inspiration and of expiration at four levels:

1. 1 cm after the confluence of the iliac veins
2. At the confluence of the renal veins
3. Immediately below the confluence of the hepatic veins
4. Immediately above the confluence of the hepatic veins (also in long axis)

At level 3 maximum and average blood velocity will be measured by Doppler provided that the angle of insonation is 60° or less.

At each level, we will compute the ratio R between the anteroposterior and lateral diameters (eccentricity) and the sectional area, calculated with the formula for the ellipse.

Statistical analysis The data obtained will be presented as mean (standard deviation). Statistical analysis will be performed with ANOVA for repeated measures and post-hoc comparisons with Student Newman Keuls test. ROC (Receiver Operating Characteristic) curves will be calculated to test the predictivity of a positive fluid load test by the aforementioned parameters; the analysis will be performed at the level at which each parameter shows the largest variations after the load test.

The a priori power analysis was performed on the primary endpoint, i.e. on changes of R in relation to IVC levels and fluid volume test with the program Gpower (17). The analysis was carried out on ANOVA with a 4 x 2 design by assuming an α error of 0.05, a power of 1-β of 0.95, and an f of 0.40, which corresponded to a large-size effect. The index f is a standardized measure of the effect size and is equal to the minimum difference considered clinically relevant divided by the standard deviation in the population. Since, the standard deviation of R was 0.1 in a previous study on healthy volunteers, an f value of 0.4 corresponded to a minimal difference of 0.04 between R values. On this basis, we obtained 112 determinations over all groups of the design, which corresponded to a sample of 14 patients (112/8=14); such value was increased by 10%, and the final sample of 16 patients was obtained.

ELIGIBILITY:
Inclusion Criteria:

* the need determined by the attending physician to perform a rapid fluid load test to guide infusions
* a condition of adequate sedation and good adaptation to mechanical ventilation
* the presence of an arterial catheter and a catheter in the pulmonary artery

Exclusion Criteria:

* obesity (BMI> 30 kg/m2)
* age <18 years
* women of childbearing age
* tricuspid insufficiency
* hemodynamically significant right ventricular failure
* bleeding from the surgical drains greater than 150 mL in the hour preceding the enrollment
* history of allergy to colloids
* administration of more than 1000 mL of hydroxyethyl starch in the last 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 16 (Estimated)
Dates: Start 2013-05; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
The eccentricity of inferior vena cava transverse sections | Baseline and after forty minutes
  The ratio R between the minimum and maximum diameters of inferior vena cava transverse sections at four different levels

SECONDARY OUTCOMES:
Blood velocity | Baseline and after forty minutes
  Maximum and average blood velocity measured immediately below the confluence of the hepatic veins by Doppler provided that the angle of insonation is 60° or less.

CONTACTS AND LOCATIONS:
Overall Officials: Franco Cavaliere, MD, Principal Investigator — Catholic University of the Sacred Heart
Locations (1):
- Catholic University of the Sacred Heart, Rome, Rome, Italy

REFERENCES:
- [Background] Kircher BJ, Himelman RB, Schiller NB. Noninvasive estimation of right atrial pressure from the inspiratory collapse of the inferior vena cava. Am J Cardiol. 1990 Aug 15;66(4):493-6. doi: 10.1016/0002-9149(90)90711-9. PMID 2386120
- [Background] Dipti A, Soucy Z, Surana A, Chandra S. Role of inferior vena cava diameter in assessment of volume status: a meta-analysis. Am J Emerg Med. 2012 Oct;30(8):1414-1419.e1. doi: 10.1016/j.ajem.2011.10.017. Epub 2012 Jan 4. PMID 22221934
- [Background] Arthur ME, Landolfo C, Wade M, Castresana MR. Inferior vena cava diameter (IVCD) measured with transesophageal echocardiography (TEE) can be used to derive the central venous pressure (CVP) in anesthetized mechanically ventilated patients. Echocardiography. 2009 Feb;26(2):140-9. doi: 10.1111/j.1540-8175.2008.00772.x. Epub 2008 Nov 24. PMID 19054047
- [Background] Lorsomradee S, Lorsomradee S, Cromheecke S, ten Broecke PW, De Hert SG. Inferior vena cava diameter and central venous pressure correlation during cardiac surgery. J Cardiothorac Vasc Anesth. 2007 Aug;21(4):492-6. doi: 10.1053/j.jvca.2006.09.009. Epub 2006 Dec 22. PMID 17678773
- [Background] Barbier C, Loubieres Y, Schmit C, Hayon J, Ricome JL, Jardin F, Vieillard-Baron A. Respiratory changes in inferior vena cava diameter are helpful in predicting fluid responsiveness in ventilated septic patients. Intensive Care Med. 2004 Sep;30(9):1740-6. doi: 10.1007/s00134-004-2259-8. Epub 2004 Mar 18. PMID 15034650
- [Background] Goldhammer E, Mesnick N, Abinader EG, Sagiv M. Dilated inferior vena cava: a common echocardiographic finding in highly trained elite athletes. J Am Soc Echocardiogr. 1999 Nov;12(11):988-93. doi: 10.1016/s0894-7317(99)70153-7. PMID 10552361
- [Background] Kimura BJ, Dalugdugan R, Gilcrease GW 3rd, Phan JN, Showalter BK, Wolfson T. The effect of breathing manner on inferior vena caval diameter. Eur J Echocardiogr. 2011 Feb;12(2):120-3. doi: 10.1093/ejechocard/jeq157. Epub 2010 Oct 27. PMID 20980326
- [Background] Ho JD, Dawes DM, Moore JC, Caroon LV, Miner JR. Effect of position and weight force on inferior vena cava diameter--implications for arrest-related death. Forensic Sci Int. 2011 Oct 10;212(1-3):256-9. doi: 10.1016/j.forsciint.2011.07.001. Epub 2011 Jul 27. PMID 21798678
- [Background] Saul T, Lewiss RE, Langsfeld A, Radeos MS, Del Rios M. Inter-rater reliability of sonographic measurements of the inferior vena cava. J Emerg Med. 2012 May;42(5):600-5. doi: 10.1016/j.jemermed.2011.05.095. Epub 2012 Jan 12. PMID 22244287
- [Background] Cavaliere F, Cina A, Biasucci D, Costa R, Soave M, Gargaruti R, Bonomo L, Proietti R. Sonographic assessment of abdominal vein dimensional and hemodynamic changes induced in human volunteers by a model of abdominal hypertension. Crit Care Med. 2011 Feb;39(2):344-8. doi: 10.1097/CCM.0b013e3181ffe0d2. PMID 21099427
- [Background] Moreno FL, Hagan AD, Holmen JR, Pryor TA, Strickland RD, Castle CH. Evaluation of size and dynamics of the inferior vena cava as an index of right-sided cardiac function. Am J Cardiol. 1984 Feb 1;53(4):579-85. doi: 10.1016/0002-9149(84)90034-1. PMID 6695787
- [Background] Willenberg T, Clemens R, Haegeli LM, Amann-Vesti B, Baumgartner I, Husmann M. The influence of abdominal pressure on lower extremity venous pressure and hemodynamics: a human in-vivo model simulating the effect of abdominal obesity. Eur J Vasc Endovasc Surg. 2011 Jun;41(6):849-55. doi: 10.1016/j.ejvs.2011.02.015. Epub 2011 Mar 16. PMID 21414818
- [Background] Murphy EH, Johnson ED, Arko FR. Evaluation of wall motion and dynamic geometry of the inferior vena cava using intravascular ultrasound: implications for future device design. J Endovasc Ther. 2008 Jun;15(3):349-55. doi: 10.1583/08-2424.1. PMID 18540710
- [Background] Murphy EH, Arko FR, Trimmer CK, Phangureh VS, Fogarty TJ, Zarins CK. Volume associated dynamic geometry and spatial orientation of the inferior vena cava. J Vasc Surg. 2009 Oct;50(4):835-42; discussion 842-3. doi: 10.1016/j.jvs.2009.05.012. Epub 2009 Aug 6. PMID 19660896